CLINICAL TRIAL: NCT05455879
Title: Impact of the Number of Doses of Antenatal Corticosteroid Therapy on the Number of Doses of Surfactants Postnatal in Preterm Infants
Brief Title: Impact of Antenatal Corticosteroid Therapy on Postnatal Surfactant Use in Preterm Infants
Acronym: CORISURF
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD0822
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2022-10

CONDITIONS: Hyaline Membrane Disease (HMD)
Keywords: Corticosteroid therapy; Surfactants; Preterm infants
MeSH Terms: conditions — Hyaline Membrane Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Impact of antenatal corticosteroid therapy on surfactants use postnatal: Intervention Description: Retrospective study on preterm infants to evaluate the impact of antenatal corticosteroid therapy on surfactants use postnatal
  Interventions: Other: Impact of antenatal corticosteroid therapy on surfactants use postnatal

INTERVENTIONS:
Other: Impact of antenatal corticosteroid therapy on surfactants use postnatal — Intervention Description: Retrospective study on preterm infants to evaluate the impact of antenatal corticosteroid therapy on surfactants use postnatal

SUMMARY:
No study has shown that two doses of corticosteroids are more effective than a single dose in lung maturation and prevention of hyaline membrane disease (HMD) The aim of this study is to assess the impact of the number of doses on the severity of HMD.

DETAILED DESCRIPTION:
Respiratory distress syndrome (RDS), formerly known as hyaline membrane disease, is a common problem in preterm infants. This disorder is caused primarily by deficiency of pulmonary surfactant in an immature lung. RDS is a major cause of morbidity and mortality in preterm infants.

Surfactant therapy has been shown to significantly reduce neonatal and infant mortality. Corticosteroids are given antenatal, and then surfactant is given, along with corticosteroids, postnatal.

A single course of corticosteroids is recommended for pregnant women between 24 weeks and 34 weeks of gestation who are at risk of preterm delivery within 7 days, including those with ruptured membranes and multiple pregnancies.

Betamethasone is recommended as the steroid of choice, to be administered in two doses of 12 mg given intramuscularly 24 hours apart.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants ≤ 37 SA
* Hospitalized in the neonatal intensive care unit between January 2018 and December 2019
* Having received at least one dose of corticosteroids antenatal

Exclusion Criteria:

* Parental Opposition
* Congenital malformations that may cause neonatal respiratory distress.

Max Age: 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm infants (≤ 37 SA), hospitalized in the neonatal intensive care unit between January 2018 and December 2019 and having received at least one dose of corticosteroids antenatal
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2022-06-20 (Actual); Primary Completion 2022-07-05 (Actual); Study Completion 2022-07-05 (Actual)

PRIMARY OUTCOMES:
Assessment of the effect of a full course of antenatal corticosteroid therapy versus a half course on the number of postnatal surfactant doses in preterm infants. | At the end of the study, an average of 2 month
  Comparison of the number of doses of surfactants administered postnatal in preterm infants who received 2 doses of antenatal corticosteroid therapy versus those who received a single dose

SECONDARY OUTCOMES:
Assessment of the influence of gestational age on the severity of hyaline membrane disease (HMD) | At the end of the study, an average of 2 month
  Radiological stage of HMD according to gestational age :
  Stage 1 : reticulo-granular appearance / borderline normal imaging of the lung, Stage 2 : diffuse reticulo-granular appearance / Visible mediastinal borders Stage 3 : global decrease in lung transparency / Bronchogram aerial / Blurred mediastinal borders Stage 4 : white lungs
Assessment of the influence of the cause of prematurity on the severity of hyaline membrane disease (HMD) | At the end of the study, an average of 2 month
  Radiological stage of HMD according to cause of prematurity :
  Stage 1 : reticulo-granular appearance / borderline normal imaging of the lung, Stage 2 : diffuse reticulo-granular appearance / Visible mediastinal borders Stage 3 : global decrease in lung transparency / Bronchogram aerial / Blurred mediastinal borders Stage 4 : white lungs
Assessment of the impact of the number of doses of antenatal corticosteroid therapy on the use of postnatal corticosteroid therapy | At the end of the study, an average of 2 month
  Prevalence of postnatal corticosteroid therapy by number of doses of antenatal corticosteroid therapy
Assessment of the impact of the number of doses of antenatal corticosteroid therapy on the prevalence of bronchopulmonary dysplasia | At the end of the study, an average of 2 month
  Prevalence of bronchopulmonary dysplasia as a function of the number of doses of antenatal corticosteroid therapy
Assessment of the impact of the number of doses of antenatal corticosteroid therapy on the severity of intraventricular hemorrhage | At the end of the study, an average of 2 month
  Stage of intraventricular hemorrhage on transfontanellar ultrasound (FET) according to the number of doses of antenatal corticosteroid therapy :
  Stage 1 : Germline or subependymal hemorrhage (SEH), Stage 2 : Ventricular hemorrhage Stage 3 : Ventriculomegaly (VM) Stage 4 : Hemorrhage in the brain parenchyma

CONTACTS AND LOCATIONS:
Overall Officials: Dr Suzanne BORRHOMEE, Principal Investigator — Hôpital NOVO
Locations (1):
- Resuscitation and neonatal medicine department - Centre Hospitalier René Dubos, Pontoise, France